CLINICAL TRIAL: NCT02916472
Title: 'Rainbow Riders': A Pilot Trial of CyberCycling to Reduce Therapeutic Side Effects and Improve Quality of Life in Adolescent and Young Adults (AYA) Diagnosed With Cancer
Brief Title: CyberCycling to Reduce Therapeutic Side Effects and Improve Quality of Life in AYA Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4Z16
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Adolescent and Young Adult Cancers
Keywords: AYA; exercise; cancer; cybercycling
MeSH Terms: conditions — Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CyberCycling - Aerobic Exercise (Experimental): 30-60 mins/week, 3 days/week supervised stationary cycling with exergaming/videogaming for 12 weeks
  Interventions: Behavioral: CyberCycling
- Control Stretching - Resistance Bands (Active Comparator): 2 days/week at home for 12 weeks
  Interventions: Behavioral: Stretching; Behavioral: Resistance Bands

INTERVENTIONS:
Behavioral: CyberCycling — All exercise training will be performed under the supervision of a qualified exercise trainer certified in Advanced Cardiac Life Support. Participants in the exercise groups will be asked to perform aerobic exercise on a stationary bike ('cybercycle') 3 days per week for 12 weeks. Exercise intensity and duration will be based on a progressive program and adapted, as needed, based on the participants' tolerability. Heart rate will be monitored throughout the exercise session and Rating of Perceived Exertion (RPE) monitored at least every 10 minutes. The target heart rate (THR) zone will be determined using the Karvonen formula.
  Other Names: stationary bikes; aerobic exercise
  Arms: CyberCycling - Aerobic Exercise
Behavioral: Stretching — Participants randomized to the control condition will receive a progressive resistance training program with TheraBands™ and a stretching program to complete at home 2 days/week for 12 weeks. The resistance band program will include upper body and lower body exercises. Participants will be provided with two different colored resistance bands (lighter colored - easier resistance; darker colored - harder resistance). Participants will start by completing 1-2 sets, 2 days/week with the easier/lighter band for the first 4 weeks, progress to 2-3 sets, 2 days/week with the easier band for the next 4 weeks; and, then, progress to 1-2 sets with the darker/harder band for the last 4 weeks. In addition, all participants in the 'control' condition will be advised to conduct upper body and lower body stretches 2 days/week. All resistance band exercises and stretches will be demonstrated to the participant by the exercise physiologist before the 12 week program begins.
  Arms: Control Stretching - Resistance Bands
Behavioral: Resistance Bands — Participants randomized to the control condition will receive a progressive resistance training program with TheraBands™ and a stretching program to complete at home 2 days/week for 12 weeks.
  The resistance band program will include upper body and lower body exercises and will be provided with two different colored resistance bands (one lighter colored for easier resistance; one darker colored for a harder resistance). Participants will start by completing 1-2 sets, 2 days/week with the easier/lighter band for the first 4 weeks, progress to 2-3 sets, 2 days/week with the easier band for the next 4 weeks; and, then, progress to 1-2 sets with the darker/harder band for the last 4 weeks. In addition, all participants in the 'control' condition will be advised to conduct upper body and lower body stretches 2 days/week. All resistance band exercises and stretches will be demonstrated to the participants by the exercise physiologist before the 12 week program begins.
  Arms: Control Stretching - Resistance Bands

SUMMARY:
Only a few clinical trials evaluating the potential benefits of exercise have been conducted in adolescents and young adults (AYA) with cancer and, no prior studies have evaluated the potential effects of 'cybercycling' (exergaming on a stationary bike) in AYA cancer survivors. Therefore, the study aims to conduct a pilot trial to determine feasibility (adherence, user acceptance) and to explore potential effects of a 'cybercycling' exercise program on fitness, body composition, quality of life, sleep and cognition.

DETAILED DESCRIPTION:
Objectives Specific Aim 1: To evaluate the feasibility (adherence; user acceptance: exercise tolerance, enjoyment and motivation) of performing an adaptive, moderate intensity, aerobic exercise program on a 'cybercycle' compared to control (stretching/resistance bands) in adolescent and young adults (AYA) with cancer.

(Exploratory) Aim 2: To explore the effects of an adaptive, moderate intensity aerobic exercise program using a 'cybercycle' compared to control (stretching/resistance bands) on changes in fitness, body composition, quality of life (QoL), fatigue, sleep and cognition.

Study Design/Overview:

This study is a randomized trial in 20 adolescent and young adult (AYA) cancer survivors (15-30 years old) which will comparing two intervention arms: 1) aerobic exercise on a 'cybercycle' (stationary cycling with exergaming/videogaming); and, 2) a stretching/resistance band 'control' condition.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed cancer
* completed primary treatment
* approved to be contacted by the treating oncologist/nurse practitioner
* meet screening criteria

Exclusion Criteria:

* patients unable to provide informed consent
* patients not available for follow-up testing
* patients with any pre-existing medical conditions that would be a contraindication to exercise.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Proportion of Patient Adherence as recorded by attendance log | Up to 12 weeks after beginning program
  Adherence rates will be summarized separately by treatment arm with proportions and exact confidence intervals. Feasibility will be defined as an adherence of greater than or equal to 80%

SECONDARY OUTCOMES:
Median change of peak pulmonary oxygen uptake (VO2Peak) | Up to 12 weeks after beginning program
  A linear mixed model will also be fit to the measures of VO2peak (baseline, EOP)
Median Tolerance of Exercise Intensity as measured by the Preference for and Tolerance of Exercise Intensity Questionnaire (PRETIE-Q) score | Up to 12 weeks after beginning program
Median Physical Activity Enjoyment Scale (PAES) score | Up to 12 weeks after beginning program
Median Flow State Scale (FSS) Score | Up to 12 weeks after beginning program
Median Exercise Motivations (EMI) Score | Up to 12 weeks after beginning program
Median total duration of each session | Up to 12 weeks after beginning program
  This is a measure of adherence
Median time in total heart rate zone (THZ) | Up to 12 weeks after beginning program
Median workload of participants while exercising | Up to 12 weeks after beginning program
Median speed in rpm of participants while exercising | Up to 12 weeks after beginning program

CONTACTS AND LOCATIONS:
Overall Officials: Nora Nock, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States